CLINICAL TRIAL: NCT05816031
Title: Effect of Ketogenic Diet on Peri-operative Complications of Right Laparoscopic Adrenalectomy in Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Mario Musella MD, Professor, Federico II University
Other Study IDs: KetoAdreno
Record Dates: First submitted 2023-04-02; First posted 2023-04-18 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Adrenalectomy; Status; Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Diet, Ketogenic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ketogenic diet: Patients scheduled to right laparoscopic adrenalectomy and belonging to the case arm, will be administered a standard 21 days ketogenic diet before surgery. Ketogenic diet is based on a standard diet plus a ketogenic product to be taken once daily for 21 days. In both groups patients will undergo abdominal ultrasound before surgery.
  Interventions: Dietary Supplement: Ketogenic diet
- No ketogenic diet: Ketogenic diet will not be prescribed to patients belonging to control group.

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Ketogenic diet administrated to obese patients planned for right laparoscopic adrenalectomy
  Groups: Ketogenic diet

SUMMARY:
Ketogenic diet is often prescribed to morbid obese patients scheduled for bariatric surgery in order to reduce liver size, thus making surgery less demanding. The study aim to investigate the possible effects of ketogenic diet on intra- and peri-operative complications of right laparoscopic adrenalectomy in obese patients; researchers will analyze intra- and peri-operative outcomes among obese patients who underwent laparoscopic right adrenalectomy, comparing the two arms with and without ketogenic diet.

DETAILED DESCRIPTION:
Ketogenic diet is often prescribed to morbid obese patients scheduled for bariatric surgery in order to reduce liver size, thus making surgery less demanding. Due to a standard trans abdominal laparoscopic right adrenalectomy is performed with the patient in left lateral position, it is necessary to retract liver in order to expose the right adrenal gland and the cava vein. It is therefore evident how a reduced size liver may allow a faster, easier and safer surgery. Finding a normal size liver is uncommon in patients presenting with a body mass index above 30 Kg/m2. According to this, patients scheduled to right laparoscopic adrenalectomy and belonging to the case arm, will be administered a standard 21 days ketogenic diet before surgery. Conversely this will not be prescribed to patients belonging to control group. Ketogenic diet is based on a standard diet plus a ketogenic product to be taken once daily for 21 days. In both groups patients will undergo abdominal ultrasound before surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 Kg/m2
* Planned for laparoscopic right adrenalectomy
* Age > 18y.o.
* No contraindications for ketogenic diet

Exclusion Criteria:

* Diabetes
* Patients requiring conversion to open surgery
* BMI < 30 Kg/m2
* Age < 18 y.o.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring laparoscopic right adrenalectomy
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Peri-operative complications | Complications occurring during surgery and within 30 days from surgery
  Pre and post-operative (within 30 days) complications of laparoscopic adrenalectomy

CONTACTS AND LOCATIONS:
Overall Officials: Mario Musella, Principal Investigator — Federico II University
Locations (1):
- Nunzio Velotti, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marescaux J, Mutter D, Wheeler MH. Laparoscopic right and left adrenalectomies. Surgical procedures. Surg Endosc. 1996 Sep;10(9):912-5. doi: 10.1007/BF00188482. PMID 8703150
- [Result] Gagner M, Lacroix A, Bolte E. Laparoscopic adrenalectomy in Cushing's syndrome and pheochromocytoma. N Engl J Med. 1992 Oct 1;327(14):1033. doi: 10.1056/NEJM199210013271417. No abstract available. PMID 1387700
- [Result] Leonetti F, Campanile FC, Coccia F, Capoccia D, Alessandroni L, Puzziello A, Coluzzi I, Silecchia G. Very low-carbohydrate ketogenic diet before bariatric surgery: prospective evaluation of a sequential diet. Obes Surg. 2015 Jan;25(1):64-71. doi: 10.1007/s11695-014-1348-1. PMID 25005809